CLINICAL TRIAL: NCT03806595
Title: A Pilot Study of Intranasal Lidocaine in Acute Management of Pediatric Migraine and Migraine-like Headache: A Randomized Controlled Trial
Brief Title: A Pilot Study of Intranasal Lidocaine in Acute Management of Pediatric Migraine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Garth Meckler, Pediatric Emergency Medicine Division Head, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H18-03801
Record Dates: First submitted 2018-11-23; First posted 2019-01-16 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Migraine in Children; Posttraumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal lidocaine (Experimental): 1mL of lidocaine 2% will be instilled in either the nostril ipsilateral to the headache or 1ml in each nostril in cases of bilateral headache.
  Interventions: Drug: Lidocaine 2% Injectable Solution
- Intranasal normal saline (Placebo Comparator): 1mL of saline 0.9% will be instilled in either the nostril ipsilateral to the headache or 1ml in each nostril in cases of bilateral headache.
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution

INTERVENTIONS:
Drug: Lidocaine 2% Injectable Solution — The Barre method of intranasal administration will be used to instil 1mL of lidocaine 2% in either the nostril ipsilateral to the headache or 1ml in each nostril in cases of bilateral headache.
  Arms: Intranasal lidocaine
Drug: Normal Saline Flush, 0.9% Injectable Solution — The Barre method of intranasal administration will be used to instil 1mL of saline 0.9% in either the nostril ipsilateral to the headache or 1ml in each nostril in cases of bilateral headache.
  Arms: Intranasal normal saline

SUMMARY:
Headaches in children are very common and are a source of significant distress for the patient and their family. Migraines are the most common headache disorder in children and are associated with episodic pain and other symptoms such as nausea and sensitivity to light and sound that can impair a child's ability to participate in daily activities and lead to missed school or parental missed work. When home treatment fails to relieve symptoms, children often seek care in the emergency department (ED) where a limited number of treatment options exist; while largely effective, these rescue treatments currently all require needle insertion of an intravenous line, take time to administer, result in prolonged ED stays, and have potential unpleasant side effects. In adult patients, a number of studies suggest that lidocaine, a local anesthetic administered intranasally, may provide relief of migraine and migraine-like headache pain in minutes. This approach has the benefit of working quickly, not requiring a needle, and having fewer side effects as the medication acts locally on nerves in the nose. Intranasal lidocaine has not yet been studied in children for this purpose. This study will compare the use of intranasal lidocaine to placebo. The goal of this pilot study is to provide information to inform the sample size calculation for the definitive randomized controlled trial that will aim to measure the efficacy of intranasal lidocaine as an analgesic option for children age 7 years and older who present to the Pediatric ED with a chief complaint of migraine or post traumatic headache with migraine-like features. Secondary objectives will be to report on the frequency and severity of rebound headache between the two treatment groups, adverse events of the study drug, as well as the impact on healthcare utilization measures.The investigators hypothesize that children receiving intranasal lidocaine will have faster and more effective pain recovery compared to children receiving placebo and will be less likely to require the standard therapy for migraine headache. Given very few side effects reported in adult studies and the relatively benign nature of those reported, the investigators do not expect any major safety concerns in the study. It is also hypothesized that intranasal lidocaine will lead to shorter ED visits, thus reducing use of staff and hospital resources and saving money for the healthcare system as a whole.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7-16 years
2. Migraine headache fulfilling Irma's criteria:

   * Headache lasting 1-72 hours with at least 4 out of 6 of the following features:

     * Moderate to severe episode of impaired daily activities
     * Focal localization of headache
     * Pulsatile description
     * Nausea or vomiting or abdominal pain
     * Photophobia, phonophobia, or avoidance of light and noise, or
     * Symptoms increasing with activity or resolving by rest.

   OR:
3. Post-traumatic headache as per ICHD-3 (beta edition) definition with migraine-like features (see above):

   A) Any headache fulfilling criteria C and D

   B) Traumatic injury to the head has occurred

   C) Headache is reported to have developed within 7 days after one of the following:

   i. The injury to the head, ii. Regaining of consciousness following the injury to the head, iii. Discontinuation of medication(s) that impair ability to sense or report headache following the injury to the head

   D) Headache persists for > 3 months after the injury to the head

   E) Not better accounted for by another ICHD-3 diagnosis
4. Verbal report of a pain score of 4 or greater on a 10 point numeric pain score (range 0-10 with increasing severity, i.e. 0 = no pain and 10 = most severe pain) after receiving first line therapy (non-narcotic analgesia) in either the out-patient or PED setting
5. Normal vital signs for age
6. Normal neurological exam (no focal deficits or abnormalities)

Exclusion Criteria:

1. Families not providing informed consent or assent, where appropriate
2. History of acute trauma or seizure in the preceding 24 hours
3. Clinical suspicion of or known intracranial pathology or underlying central nervous system disease
4. Headache associated with fever or meningismus
5. Known allergy/sensitivity to lidocaine

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change in migraine pain | Pain scores will be measured at 30 and 60 minutes post intranasal administration of either the study drug or placebo.
  The primary outcome measure will be the proportion of subjects with numeric pain scores of < 4 out of 10 on a verbal rating scale (range 0 -10 with increasing severity, i.e. 0 = no pain and 10 = most severe pain).Treatment success is defined as a score of 3 or less at the two time points. This will be recorded for each patient during the study timeframe, until study completion.

SECONDARY OUTCOMES:
Rebound headache | Pain scores will be recorded at 60 minutes, 24 hours, and within 48-72 hours post intranasal therapy.
  Proportion of patients with rebound headache (i.e. headache with pain score of greater than or equal to 4 out of 10 on a verbal rating scale; range 0 -10 with increasing severity, i.e. 0 = no pain and 10 = most severe pain). This will be recorded for each patient at the visit of interest during the study timeframe, until study completion.
Emergency department length of stay | The emergency department length of stay will be ascertained from the medical record within 24 hours of the participant's visit.
  Number of hours in the Emergency Department from time of registration to time of discharge or admission to hospital for each subject.
Proportion of participants discharged vs. admitted from the emergency department (emergency department disposition) | Disposition will be ascertained from the medical record within 24 hours of the participant's ED visit.
  Disposition of the patient from the emergency department for the visit of interest only, i.e. discharge home, hospital admission. This will be recorded for each patient during the study timeframe, until study completion.
Proportion of participants with a return visit to the emergency department within 72 hours of discharge. | Within 3 days from index visit.
  Returns to the emergency department for similar complaints of migraine headache or posttraumatic headache with migraine like features.

CONTACTS AND LOCATIONS:
Overall Officials: Garth Meckler, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No